CLINICAL TRIAL: NCT05742633
Title: Comparative Effect of Active Release Technique Versus Self-myofascial Release in Improving Piriformis Syndrome. A Randomized Controlled Trial
Brief Title: Comparative Effect of Active Release Technique Versus Self-myofascial Release in Improving Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ramshaakbar20
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received Active release technique (ART)
  Interventions: Other: Active release technique
- Group B (Other): Group B received self-myofascial release (SMFR)
  Interventions: Other: Self-myofascial release

INTERVENTIONS:
Other: Active release technique — Active Release Technique was applied to patient in prone lying, knee flexed at 90. The therapist placed his elbow tip on taut band of piriformis and direct pressure applied, patient wias then asked to do internal rotation of hip, in order to achieve lengthening of the muscle. This was repeated 5-7 times.
  A total of 18 sessions was given over a period of 6 weeks (3 sessions per week)
  Arms: Group A
Other: Self-myofascial release — Patient position in prone lying Therapist was standing beside the patient at the waistline, working on the contralateral side.
  Piriformis muscle was located by an imaginary line drawn between the midpoint of the lateral aspect of the sacrum and the greater trochanter. A contact was established in the gluteal area about 3 cm from the sacrum. Patent was guided to use a foam roller followed by a massage ball.
  A total of 18 sessions were given over a period of 6 weeks (3 sessions per week)
  Arms: Group B

SUMMARY:
The goal of this Randomized controlled trial is to examine comparative effect of active release technique versus self-myofascial release in improving piriformis syndrome. The main question it aims to answer is:

• To compare the effects of Active release technique (ART) and Self-Myofascial release (SMFR) on pain intensity, hip internal rotation and functional disability in patients with piriformis syndrome.

Participants will be a given consent form and after subjects read and sign the informed consent, they would be included in study according to eligibility criteria. 2 groups would be included in study, Active release technique will be applied on group A by the physiotherapist and self-myofascial release will be applied on group B by the patients themselves through the use of foam-rollers and massage ball to compare the results of both these techniques on reducing pain, improving range and functional disability among individuals with piriformis syndrome. We will measure outcome through different outcome measure tools.

DETAILED DESCRIPTION:
Piriformis is a key internal rotator of the hip which develops muscular imbalance due to overuse and pressure. There are various disabling conditions caused due to a simple tightness of Piriformis muscle like low back pain, sciatic nerve pain through muscle hypertrophy or a nearby anomaly due to its anatomically closeness to the sciatic nerve, pain and aesthesia in hip, thigh, calf and foot are symptoms that commonly occur in Piriformis syndrome. Piriformis syndrome is defined as a peripheral neuritis of the branches of the sciatic nerve caused by an abnormal condition of the piriformis muscle (PM), such as an injured or irritated muscle.

MFR technique involves application of a low load-long duration stretch to the myofascial complex which intends to restore the optimal length, decrease pain and improve functional mobility of the muscle. A special technique within MFR is self-myofascial release (SMFR), performed by the patient independently, instead of by a therapist. This technique utilizes the patient's body mass and special tools such as massage balls or foam rollers to apply pressure and stretch the restricted soft tissue. Active Release Techniques (ART) are a soft tissue method that focuses on relieving tissue tension via the removal of fibrosis/adhesions which can develop in tissues as a result of overload due to repetitive use.

Active release technique will be applied on group A by the physiotherapist and self-myofascial release will be applied on group B by the patients themselves through the use of foam-rollers and massage ball to compare the results of both these techniques on reducing pain, improving range and functional disability among individuals with piriformis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years
* males and females
* Pain more than 1 month.
* Piriformis syndrome diagnosed through screening tests (FAIR test, Beatty test, Freiberg test, Sign of Pace)
* A score ≥8 on a 12-point Clinical scoring system for diagnosis of piriformis syndrome

Exclusion Criteria:

* Inflammation, malignancy, arthritis, active infection, post-partum or pregnant females and post-op patients, any deformity.
* Leg pain due to causes other than piriformis syndrome
* Any traumatic History.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Likert pain scale (change is being assessed) | Change from Baseline at 6 weeks
  Pain intensity is principally assessed using rating scales such as the 11-point Likert scale. In general, frequent pain assessments are serially correlated and underdispersed. The aim of this investigation was to develop population models adapted to fit the 11-point pain scale.
Lower extremity functional scale (change is being assessed) | Change from Baseline at 6 weeks
  The lower extremity functional scale (LEFS) is a valid patient-rated outcome measure (PROM) for the measurement of lower extremity function.
  The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.
Range of Motion by Goniometer (change is being assessed) | Change from Baseline range of motion at 6 weeks
  Range of straight leg raise (SLR) and Internal rotation range would be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Akbar, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan